CLINICAL TRIAL: NCT01268618
Title: A Double-blind, Randomized, Placebo-controlled, Dual-center Study on the Effect of Healthy Trinity (Retail Label)/Trenev Trio (Professional Label) on Symptoms of Diarrhea-predominant Irritable Bowel Syndrome (IBS-D) and Functional Dyspepsia
Brief Title: Trenev Trio/Healthy Trinity for Symptoms of Diarrhea-predominant Irritable Bowel Syndrome (IBS) and Functional Dyspepsia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sprim Advanced Life Sciences (Other)
Responsible Party: Larry Miller, PhD, Sprim Advanced Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-SUS-05-NAT-01
Record Dates: First submitted 2010-12-28; First posted 2010-12-31 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: IBS-D and Functional Dyspepsia
Keywords: IBS; Diarrhea; Dyspepsia
MeSH Terms: conditions — Diarrhea; Dyspepsia | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Experimental)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 2 capsules, 3x/day capsules of Healthy Trinity (retail label)/Trenev Trio (professional label), for a total daily dose of:
  1. Lactobacillus acidophilus NAS, 30 billion CFU
  2. Bifidobacterium bifidum Malyoth, 120 billion CFU
  3. Lactobacillus delbrueckii subspecies bulgaricus LB-51, 30 billion CFU
  Arms: Probiotic
Dietary Supplement: Placebo — 2 capsules, 3x/day placebo capsules
  Arms: Placebo

SUMMARY:
Primary Objective:

• To confirm the efficacy of the probiotic product Healthy Trinity (retail label)/Trenev Trio (professional label) in the improvement of symptoms in adult patients with diarrhea-predominant irritable bowel syndrome (IBS-D) and functional dyspepsia

Secondary Objective:

• To confirm the safety of the probiotic product Healthy Trinity (retail label)/Trenev Trio (professional label) in adult patients with IBS-D and functional dyspepsia

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years
2. Diagnosed with IBS-D including: a) weekly average of worst abdominal pain in the last 24 hours of ≥3 on a 0-10 scale, and b) weekly average of Bristol Stool form of ≥6 on a 1-7 scale
3. Diagnosed with functional dyspepsia defined as presence of at least one of the following symptoms: bothersome postprandial fullness, early satiation, epigastric pain, or epigastric burning AND no evidence of structural disease that is likely to explain the symptoms
4. History of IBS-D and dyspepsia symptoms for at least 12 weeks
5. Agree to use contraception throughout study period, unless postmenopausal or surgically sterile (females only)
6. Able to understand the nature and purpose of the study including potential risks and side effects
7. Willing to consent to study participation and to comply with study requirements
8. Successful completion of 2-week placebo-only run-in period, defined as ≥90% product compliance and completion of required questionnaires

Exclusion Criteria:

1. Major gastrointestinal complication, e.g. Crohn's disease or ulcer
2. Prior abdominal surgery with the exception of hernia repair and appendectomy
3. Subjects over 60 years who have not had a sigmoidoscopy or colonoscopy in the past 10 years
4. Clinically significant systemic disease
5. Life expectancy < 6 months
6. Pregnant female or breastfeeding
7. Lactose intolerance
8. Immunodeficient subjects
9. Anti-psychotic medication within the prior 3 months or major psychiatric disorder within the past 2 years
10. Systemic steroids within the prior month
11. Current treatment with nasogastric tube, ostomy, or parenteral nutrition
12. Use of proton pump inhibitors
13. Eating disorder
14. Recent (< 2 weeks) antibiotic administration
15. History of alcohol, drug, or medication abuse
16. Daily consumption of probiotics, fermented milk, and/or yogurt
17. Known allergies to any substance in the study product
18. Participation in another study with any investigational product within 3 months of screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Abdominal pain severity | 8 weeks
Stool consistency (Bristol Stool Chart) | 8 weeks
Dyspepsia Symptom Severity Index (DSSI) | 8 weeks

SECONDARY OUTCOMES:
Proportion of subjects with 1 or more adverse events | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Duane Wombolt, MD, Principal Investigator — Clinical Research Associates of Tidewater; David Wyatt, MD, Principal Investigator — In-Quest Medical Research, LLC
Locations (2):
- United States (2):
  - In-Quest Medical Research, LLC, Duluth, Georgia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia